CLINICAL TRIAL: NCT06833268
Title: Real-world Outcomes of Patients With HER2-positive (HER2+) Metastatic Breast Cancer (mBC) After Treatment With Trastuzumab Deruxtecan (T-DXd) in the United States
Brief Title: Real-world Outcomes of Patients With HER2+ Metastatic Breast Cancer After Treatment With Trastuzumab Deruxtecan
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: U31402-0010-NIS-MA
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: HER2-positive Breast Cancer
Keywords: HER2-positive breast cancer; Real-world outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HER2-positive breast cancer: Patients diagnosed with HER2-positive metastatic breast cancer who initiated a subsequent LOT after the initial T-DXd-containing LOT in the metastatic setting.
  Interventions: Other: No drug

INTERVENTIONS:
Other: No drug — This is an non-interventional, observational study. No drug will be provided or administered as part of this protocol.

SUMMARY:
This study will explore treatment patterns and clinical outcomes using the US-based Flatiron Health database to describe patients with HER2+ mBC who were previously treated with T-DXd to better characterize this population and inform internal decision making in this rapidly changing therapeutic landscape.

DETAILED DESCRIPTION:
This study will utilize a longitudinal, demographically and geographically diverse database derived from Electronic Health Record data. No study medication will be supplied or administered for this protocol. The primary research objective is to describe the real-world progression-free survival (rwPFS) in HER2+ mBC patients who initiated a subsequent line of therapy (LOT) after a T-DXd-containing LOT in the metastatic setting.

Secondary research objectives include describing the real-world overall survival (rwOS), patient demographics and clinical characteristics, real-world time to next treatment (rwTTNT), and real-world time to treatment discontinuation (rwTTD) in HER2+ mBC patients who initiated a subsequent LOT after a T-DXd-containing LOT in the metastatic setting. Treatment patterns and sequencing in HER2+ mBC patients for subsequent LOTs following initial treatment with T-DXd will also be assessed.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all the inclusion criteria below to be included in the study population:

1. Patients with evidence of stage IV or recurrent mBC with a metastatic diagnosis date on or after January 1, 2011.
2. Patients aged ≥18 years old at mBC diagnosis date.
3. Patients with ≥1 T-DXd-containing LOT in the metastatic setting.
4. Patients with evidence of a subsequent LOT following the first T-DXd-containing LOT in the metastatic setting. The LOT subsequent to the first T-DXd-containing LOT in the metastatic setting will be the index LOT. Index date will be the index LOT start date.
5. Patients whose closest HER2 test result (defined as immunohistochemistry [IHC] 3+ or in situ hybridization [ISH]+) recorded prior to or on the index date was a HER2+ test result.
6. Patients with index date occurring at least 90 days prior to end of study period (March 31st, 2024).

Exclusion Criteria No exclusion criteria will be imposed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults in the Flatiron mBC EDM who were diagnosed with HER2+ mBC during the study period and initiated a subsequent LOT after the initial T-DXd-containing LOT in the metastatic setting.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Real-world Progression-free Survival (rwPFS) | Index date (index LOT start date) to date of earliest disease progression >14 days after the index date or date of death, whichever occurs first, up to approximately 13 years 3 months
  rwPFS is defined as the interval in months between the index date until the first evidence of progression or death as documented by Flatiron.

SECONDARY OUTCOMES:
Real-world Time to Next Treatment (rwTTNT) | Index date (index LOT start date) to next LOT start date or, in the absence of next LOT, death, whichever occurs first, up to approximately 13 years 3 months
  rwTTNT is defined as the time in months between index date and initiation of next LOT, or death, whichever occurs first.
Real-world Time to Treatment Discontinuation (rwTTD) | Index date (index LOT start date) to date treatment is discontinued, up to approximately 13 years 3 months
  rwTTD is defined as the time in months between index date and date of treatment discontinuation or death, whichever occurs first.
Treatment Patterns by Type of Line of Therapy | Index date (index LOT start date) to end of study period, up to approximately 13 years 3 months
  Treatment patterns will be described by LOT (monotherapy, combination therapy, and treatment sequence).

CONTACTS AND LOCATIONS:
Overall Officials: Project Manager, Study Director — Daiichi Sankyo
Locations (1):
- Flatiron Health, Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No